CLINICAL TRIAL: NCT04680013
Title: Genetic Studies in Familial Dementia
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Case Western Reserve University (Other); Columbia University (Other); Wake Forest University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Margaret Pericak-Vance, Professor, University of Miami
Other Study IDs: 20070307; RF1AG054080 (NIH); RF1AG054074 (NIH); U01AG052410 (NIH)
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Dementia of Alzheimer Type; Alzheimer Disease, Late Onset; Alzheimer Disease, Early Onset; Mild Cognitive Impairment; Dementia
Keywords: Memory loss
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Memory Disorders

STUDY DESIGN:
Biospecimen Retention: Approximately 40 ml of whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cognitive Control: Participants in this group are cognitively intact.
- Mild Cognitive Impairment: Participants in this group have mild cognitive impairment.
- Dementia Group: Participants in this group have dementia.

SUMMARY:
The purpose of this study is to identify genetic factors that contribute to or cause dementia (loss of memory) and related disorders across all ages and ethnic groups. This includes a number of neurological diseases such as early and late-onset Alzheimer disease, mild cognitive impairment, and other dementias.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older
2. Patients diagnosed with dementia, their family members and unrelated healthy controls without dementia.

Exclusion Criteria:

1. Individuals with competing diagnosis such as: Amyotrophic lateral sclerosis, Frontotemporal lobar degeneration, Multiple system atrophy, Corticobasal degeneration, Progressive Supranuclear Palsy, Huntington's disease, traumatic brain injury, drug or alcohol abuse, or schizophrenia, etc. (unless family members of a dementia affected individual).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of older individuals affected by dementia, mild cognitive impairment, cognitive controls, or their family members. Ascertainment is across both males and females, and all race-ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 4884 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Correlation between genetic factors and Alzheimer disease, dementia, and related phenotypes. | 5 years
  Genetic factors will be measured through genome-wide genotyping arrays and/or whole-genome sequencing, and then correlated with Alzheimer disease and related phenotypes, such as cognitive impairment, functional impairment, and relevant biomarkers.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Pericak-Vance, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be shared via government required repositories and with our collaborators. Data are coded, with no personally identifiable information included. Data shared include the genomic data (array data, sequence data, APOE genotyping results, etc), phenotype data (case/control status, age of onset, etc), and basic demographic information (sex, race/ethnicity data if available, etc).
  The NIH Genomic Data Sharing Policy (GDS Policy) took effect on January 25th, 2015. This necessitates that we send coded data and samples to the National Institute on Aging Genetics of Alzheimer's Disease (NIAGADS)l; in some cases materials derived from participants (blood or DNA) may be stored at the National Cell Repository for Alzheimer's Disease (NCRAD).
  We may share deidentified genomic and phenotypic data with collaborators at other sites in order the accomplish the scientific aims of the study. Such research is performed with the approval of the local internal review boards.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This study adheres to the NIA Alzheimer Disease Genomics Data Sharing Plan (https://www.nia.nih.gov/research/dn/alzheimers-disease-genomics-sharing-plan). As such, genomic data will be deposited in NIH/NIA data repositories (www.niagads.org). For genomic data, this typically happens within a year of data generation, or upon publication in scientific journals (whichever is sooner). Basic phenotypic data (affection status, age of onset, sex, family structure if applicable, etc) are deposited with the genomic data. More detailed phenotypic data (cognitive data, biomarker, etc) will be made available upon publication. Data dictionaries for primary data (genomic data and basic phenotypic data) will be available with the deposition of data into the NIH/NIA data repositories (www.niagads.org). Additional supporting documentation (analysis plans, study protocols, etc) is typically described in detail upon publication of results in peer reviewed literature.
Access Criteria: This study adheres to the NIA Alzheimer disease Genomics Data Sharing Plan (https://www.nia.nih.gov/research/dn/alzheimers-disease-genomics-sharing-plan). As part of this plan data distribution agreements are required before recipients receive any data from this study. The primary requirements for the DDA include language ensuring that (1) data are not transferred to others beyond the initial recipient, (2) no attempt will be made to identify participants, (3) any results or data generated as part of the study will be shared back to NIA/NIAGADS. See the NIA Data Distribution Agreement for more details (https://www.niagads.org/sites/all/public_files/NIAGADS-DDA.pdf).
URL: https://www.nia.nih.gov/research/dn/alzheimers-disease-genomics-sharing-plan

REFERENCES:
- See also: NIA Genomics of Alzheimer Disease Storage site — http://www.niagads.org